CLINICAL TRIAL: NCT07373288
Title: HOXB7 and Linked Tissue and Blood Biomarkers in the Lungs of Patients With Pulmonary Fibrosis
Acronym: HOGWARTS
Status: Recruiting | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Roberto Tonelli, Principal investigator, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio20
Record Dates: First submitted 2025-04-24; First posted 2026-01-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Fibrosis, Pulmonary
Keywords: Idiopathic pulmonary fiborsis; Criobiopsy; Lung proteomic; Lung transcriptomic
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients undergoing surgical lung biopsy/criobiopsy for clinical purpose in the diagnostic work-up of ILD.
  Interventions: Procedure: Biopsy
- Controls: Patients undergoing lung lobectomy for lung cancer suspicion.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — This is a non-therapeutic, observational sampling study. Procedures include:
  Lung tissue sampling via:
  Surgical biopsy Transbronchial cryobiopsy Explanted lungs from transplant patients Blood sampling for exosome analysis

SUMMARY:
This pilot, multicenter, interventional study investigates the expression of HOXB7 and its associated molecular pathway in lung tissue and blood-derived exosomes from patients with pulmonary fibrosis (PF), including idiopathic pulmonary fibrosis (IPF). Using RNA sequencing (RNA-Seq) and proteomic analysis via mass spectrometry (MS), the study aims to identify tissue and circulating biomarkers associated with fibrosis progression. The study compares different biopsy techniques (surgical vs. transbronchial cryobiopsy) and also includes a control group of patients undergoing lung resection for non-fibrotic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 with clinical suspicion of pulmonary fibrosis
* Availability of fresh lung tissue from biopsy or lung explant
* Signed informed consent for research use of biological material and data

Exclusion Criteria:

- Refusal to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients aged 18 to 80 years with clinical suspicion of pulmonary fibrosis, admitted to the Center for Rare Lung Diseases (MaRP) at the University Hospital of Modena (AOU Policlinico di Modena), or to collaborating centers.
  An additional control group will consist of adult patients undergoing lung resection for reasons unrelated to fibrotic interstitial lung diseases (e.g., neoplastic conditions), enrolled at the same institutions.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
HOXB7 Expression | Baseline
  HOXB7 gene and protein expression in lung biopsy samples

SECONDARY OUTCOMES:
Assessment of RNA content | Baseline
  Comparison of RNA content between surgical and cryobiopsy samples Identification of HOXB7-positive LR-MSCs from fresh biopsy tissue Exosomal biomarkers associated with HOXB7 expression in serum Feasibility and yield of RNA-Seq and proteomics from fresh vs. snap-frozen tissues
Assessment of proteins content | Baseline
  Comparison of protein content between surgical and cryobiopsy samples

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico di Modena, Modena, Italy